CLINICAL TRIAL: NCT05958511
Title: Assessment of Risk Factors and Outcome of Thrombocytopenia in Intensive Care Unit Patients in Assiut Pediatric University Hospital
Brief Title: Assessment of Risk Factors and Outcome of Thrombocytopenia in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Metwli Hammam, Principal Investigator, Assiut University
Other Study IDs: Thrombocytopenia
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The many comorbidities in the severely ill patient also make thrombocytopenia very common (∼ 40%) in intensive care unit patients. The risk of bleeding is high with severe thrombocytopenia and is enhanced in intensive care patients with mild or moderately low platelet counts when additional factors are present that interfere with normal hemostatic mechanisms (eg, platelet function defects, hyperfibrinolysis, invasive procedures, or catheters).

DETAILED DESCRIPTION:
The many comorbidities in the severely ill patient also make thrombocytopenia very common (∼ 40%) in intensive care unit patients. The risk of bleeding is high with severe thrombocytopenia and is enhanced in intensive care patients with mild or moderately low platelet counts when additional factors are present that interfere with normal hemostatic mechanisms (eg, platelet function defects, hyperfibrinolysis, invasive procedures, or catheters). Even if not associated with bleeding, low platelet counts often influence patient management and may prompt physicians to withhold or delay necessary invasive interventions, reduce the intensity of anticoagulation, order prophylactic platelet transfusion, or change anticoagulants due to fear of heparin-induced thrombocytopenia.

The many comorbidities in the severely ill patient also affect platelet homeostasis, and, consequently, thrombocytopenia is very common in critically ill patients treated in the intensive care unit (ICU). Thrombocytopenia is usually defined as a platelet count of < 150 × 109/L, whereas severe thrombocytopenia is considered as platelet counts < 50 × 109/L. Thrombocytopenia has six major mechanisms, and it can be induced by hemodilution, increased platelet consumption (both are very common in the ICU after tissue trauma, bleeding, and disseminated intravascular coagulopathy [DIC]), increased platelet destruction (ie, immune mechanisms), decreased platelet production, increased platelet sequestration, or by the laboratory artefact of pseudothrombocytopenia .

ELIGIBILITY:
Inclusion Criteria:

* Children and infants aged one month to 18 years admitted to the ICU in period from August 2023 to August 2024 and developed thrombocytopenia documented in laboratory investigation done in PICU.

Exclusion Criteria:

* patients older than 18 years
* Patients diagnosed with congenital thrombocytopenia (TAR syndrome...etc)

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 130 Children and infants aged one month to 18 years admitted to the ICU in period from August 2023 to August 2024 and developed thrombocytopenia documented in laboratory investigation done in PICU.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Identify the prevalence thrombocytopenia. | Baseline
  The study is aimed to identify the prevalence of thrombocytopenia in patients admitted to pediatric intensive care unit.
Identify the risk factors of thrombocytopenia | Baseline
  The study is aimed to identify the risk factors of thrombocytopenia in patients admitted to pediatric intensive care unit.
Identify the outcome of thrombocytopenia | Baseline
  The study is aimed to identify the outcome of thrombocytopenia in patients admitted to pediatric intensive care unit.